CLINICAL TRIAL: NCT01782768
Title: Comparative Effects of Noninvasive Proportional Assist and Pressure Support Ventilation on Neural Respiratory Drive in Recovering Acute Exacerbation of Chronic Obstructive Pulmonary Disease(AECOPD) Patients
Brief Title: Comparative Effects of Different Noninvasive Ventilation Mode on Neural Respiratory Drive in Recovering AECOPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Zhang Jianheng, zhang jianheng, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: zjianheng
Record Dates: First submitted 2013-01-19; First posted 2013-02-04 (Estimated); Last update posted 2016-12-06 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Neural respiratory drive in different level of NPPV
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Effect of different NPPV mode on NRD (Experimental): 13 hypercapnic recovering AECOPD patients were placed on different mode of noninvasive positive pressure ventilation(NPPV,such as the PAV or PSV mode) randomly.For each mode, three levels (PA-, PA, PA+or PS-, PS, PS+), ) of support were applied.PS and PA are set for the patient's comfort . On the basis of these two levels, 25% increase and reduction assisted level of pressure were set both for PS and PA (PA-, PA+or PS-, PS+). At each level, the patients were ventilated at least 20 minutes until the breathing was stable.
  Interventions: Device: noninvasive positive pressure ventilation

INTERVENTIONS:
Device: noninvasive positive pressure ventilation — the assisted level of the noninvasive proportional assist(PAV) and pressure support ventilation(PSV) on Neural respiratory drive(NRD) in recovering patients with acute exacerbation of chronic obstructive pulmonary disease

SUMMARY:
Background: The efﬁciency of Neural respiratory drive (NRD)expressed by a ratio of ventilation to the diaphragm electromyogram (EMGdi) decreases in patients with COPD .Improving the neural respiratory drive efficiency of COPD will help to relieve the clinical symptom and make the patients feel comfort.Noninvasive positive pressure ventilation(NPPV)is a good treatment to AECOPD patients.It is unknown the effects of different mode of noninvasive positive pressure ventilation(NPPV) such as proportional assist ventilation (PAV) and pressure-support ventilation (PSV) on the efﬁciency of Neural drive of AECOPD and which mode benefit the patients more.

Objective: To compare the short-term effects of mask pressure support ventilation (PSV) and proportional assist ventilation (PAV) on Neural respiratory drive in recovering patients of AECOPD

DETAILED DESCRIPTION:
Methods: After the baseline data of spontaneous breathing was collected, 20 hypercapnic recovering AECOPD patients were placed on different mode of noninvasive positive pressure ventilation(NPPV, such as the PAV or PSV mode) randomly. For each mode, three levels (PA-, PA, PA+or PS-, PS, PS+), ) of support were applied.PS and PA are set for the patient's comfort . On the basis of these two levels, 25% increase and reduction assisted level of pressure were set both for PS and PA (PA-, PA+or PS-, PS+). At each level, the patients were ventilated at least 20 minutes until the breathing was stable. The respiratory frequency (RR), tidal volume (VT), transdiaphragmatic pressure (pdi) the pressure-time product (PTP) and root-mean-square(RMS) of EMGdi were calculated. Esophageal and gastric balloon-catheters were used to detect the intra-thoracic and abdominal pressure. Airway pressure was also measured simultaneously. EMGdi was recorded from a multipair esophageal electrode .During ventilation Airflow and ventilation were measured with pneumotachograph.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of the COPD (Chronic Obstructive Pulmonary Disease) the COPD patients were all in stable condition during recovery from acute exacerbation.

Exclusion Criteria:

* severe Cardiovascular disease
* Pneumonia
* neuromuscular and chest wall deformity
* Respiratory arrest
* Cardiovascular instability (hypotension, arrhythmias, myocardial infarction)
* Change in mental status; uncooperative patient
* High aspiration risk
* Viscous or copious secretions
* Recent facial or gastroesophageal surgery
* Craniofacial trauma
* Fixed nasopharyngeal abnormalities
* Burns
* Extreme obesity

Ages: 50 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-01; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
change of the Neural respiratory drive | 15-20 minute
  In recent studies, The efficiency of neural respiratory drive(NRD) as expressed as a ratio of minute ventilation to diaphragm electromyogram (EMGdi) in patients with COPD is lower than that in healthy subject, suggesting that, to achieve the same minute ventilatory volume, a higher neural drive is required for patients with COPD than for healthy individuals.Furthermore,levels of neural respiratory drive were related to disease severity and dyspnea.Improving the neural respiratory drive efficiency of COPD will help to relieve the clinical symptom and make the patients feel comfort. Because dyspnea relates to respiratory effort.Neural respiratory drive(NRD) and its efficiency as expressed by a ratio of ventilation to the diaphragm electromyogram(EMGdi)may be a good tool to evaluate treatment benefits in Patients with COPD.This study want to investigate the effect of noninvasive positive pressure ventilation(NPPV)on the Neural respiratory drive of COPD patients

SECONDARY OUTCOMES:
change of the pressure-time product(PTP) | 15-20 minute
  The pressure-time product(PTP)means inspiratory effort of the inspiratory muscle In COPD lung mechanical abnormality including airflow obstruction and dynamic hyperinflation and intrinsic positive end-expiratory pressure increase the work load of the respiratory muscles,which will lead to higher inspiratory work. As a result,The efficiency of neural respiratory drive as expressed as a ratio of minute ventilation to diaphragm electromyogram (EMGdi) in patients with COPD is lower than that in healthy subject.This study want to investigate the effect of noninvasive positive pressure ventilation(NPPV)on the inspiratory muscle load of the COPD patients

CONTACTS AND LOCATIONS:
Overall Officials: rong chang chen, professor, Study Director — TheFirst Affiliated Hospital Of Guangzhou Medical Collage
Locations (1):
- TheFirst Affiliated Hospital Of Guangzhou Medical Collage, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Zhang J, Luo Q, Chen R. Patient-Ventilator Interaction With Noninvasive Proportional Assist Ventilation in Subjects With COPD. Respir Care. 2020 Jan;65(1):45-52. doi: 10.4187/respcare.06430. Epub 2019 Sep 24. PMID 31551283